CLINICAL TRIAL: NCT07028151
Title: Comparison of the Effects of Classical Massage and Conventional Treatment Methods in Phone Addicted Bruxist Patients
Acronym: Bruxism
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Miraç Sezer, lecturer, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-SBB-0226
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Bruxism; Physiotherapy; Orafacial Pain
Keywords: Bruxism; Physical Therapy; Massage; TENS; Ultrasound; Pain
MeSH Terms: conditions — Bruxism; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Thirty patients with bruxism were randomly divided into as Manual Therapy Group (15) and Conventional Treatment Group (15).
Who Masked: Outcomes Assessor
Masking Description: To ensure blinding, baseline and final outcome measurements were performed by researchers other than the physiotherapist performing manual therapy and Conventional Treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy (Experimental): Participants who meet the inclusion criteria will be evaluated after providing written informed consent and will receive 10 sessions of approximately 40 minutes of classical face and neck massage
  Interventions: Other: manual therapy
- Conventional Therapy (Experimental): Participants who meet the inclusion criteria will be evaluated after providing written informed consent and will commence the treatment sessions. Each session will consist of sequential applications of infrared therapy, ultrasound, and transcutaneous electrical nerve stimulation (TENS). The sessions, lasting approximately 40 minutes each, will be conducted over a total of 10 days
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: manual therapy — Participants who meet the inclusion criteria will be evaluated following the acquisition of written informed consent. Treatment will be administered with participants in the supine position. Initially, soft tissue mobilization will be applied to the cervical extensor muscle group, followed by gentle cervical vertebral traction. Subsequently, a classical facial massage will be performed. The massage will include the suprahyoid muscles and the medial pterygoid. Intramuscular stretching and friction massage techniques will be applied to the masseter and anterior temporalis muscles. Each session will last approximately 40 minutes and will be conducted over a total of 10 sessions."
  Arms: Manual Therapy
Other: Conventional Therapy — Participants who meet the inclusion criteria will be evaluated after providing written informed consent. Treatment will be administered with participants in the supine position. Protective goggles will be placed on the participants' eyes prior to the infrared therapy application. Following 20 minutes of infrared treatment, ultrasound (1 MHz) will be applied to the masseter muscle using the full-contact method for 3 minutes. Finally, transcutaneous electrical nerve stimulation (TENS) will be applied to the masseter and anterior temporalis muscles for 15 to 20 minutes. Each session will last approximately 40 minutes and will be conducted over a total of 10 sessions.
  Arms: Conventional Therapy

SUMMARY:
Bruxism, defined as the involuntary clenching or grinding of teeth during sleep or wakefulness, is a common condition with multifactorial etiology. It can lead to various complications including temporomandibular joint (TMJ) pain, masticatory muscle hypertrophy, dental wear, headaches, and postural dysfunction. Although its underlying causes remain unclear, stress, poor sleep quality, postural problems, and excessive smartphone use have been identified as potential contributing factors.

Recent studies suggest a significant relationship between bruxism and psychological as well as behavioral variables such as stress levels, screen time, and physical inactivity. University students, due to academic pressure and lifestyle habits, may be particularly vulnerable.

This study aims to investigate the relationship between bruxism and smartphone addiction, sleep quality, and perceived stress among associate degree students at Bartın University. By identifying these associations, the study seeks to contribute to preventive strategies and promote awareness of bruxism-related risk factors in young adults.

DETAILED DESCRIPTION:
Bruxism is a common multidisciplinary condition characterized by involuntary teeth clenching or grinding that occurs during sleep or wakefulness. Although bruxism episodes are typically short in duration, they can lead to significant complications involving the masticatory muscles and postural system, including temporomandibular joint (TMJ) pain and dysfunction, headaches, dental wear, hypersensitivity, tooth pain, hypertrophy of the masticatory muscles, implant fractures, and joint sounds. While its etiology is not fully understood, bruxism is believed to be multifactorial. Studies suggest that a lifestyle characterized by chronic stress and smartphone dependency may trigger or exacerbate bruxism. Additionally, poor sleep quality and postural abnormalities have been shown to influence both bruxism and emotional stress levels, while low levels of physical activity may further impair sleep and increase stress.

The aim of this study is to improve symptoms and enhance the quality of life in individuals with smartphone addiction and bruxism complaints through the application of different physiotherapy interventions.

Following the approval of the Ethics Committee of Bartın University Vocational School of Health Services, the study will be initiated. Data collection will take place between May 2025 and September 2025. A total of 30 university students diagnosed with bruxism and enrolled at Bartın University will be included in the study. Participants will be randomly assigned using a coin toss method into two groups: a massage group (MG, n=15) receiving classical face and neck massage, and a treatment group (TG, n=15) undergoing a conventional physiotherapy program including transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound, and infrared heat therapy.

After obtaining written informed consent from eligible participants, all assessments will be conducted in the same order by a blinded assessor. Following baseline evaluations, participants will undergo 10 sessions of their respective treatment protocols, each lasting approximately 40 minutes. The MG will receive classical massage, while the TG will receive TENS, ultrasound, and infrared therapy. After completion of the intervention sessions, post-treatment evaluations will be carried out by the same assessor, and the data will be subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

Volunteer students aged between 18-27

Having at least two clinical signs of bruxism Abnormal tooth wear on the occlusal surfaces of the teeth Abfraction Gingival recession and/or cervical defect Tongue indentations or damage to the inside of the cheek Tense facial and jaw muscles, muscle sensitivity, and masseteric hypertrophy upon bidigital palpation

Exclusion Criteria:

* Characterized by a neurological disease,
* Botulinum toxin injections into the masticatory muscles in the last year,
* Using antidepressant-type medications that will affect the central nervous system,
* Receiving occlusal splint treatment,

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Level | From baseline to the end of treatment at 10 days
  A visual analog scale (VAS) will be used to assess the severity of pain associated with bruxism. The patient will be asked to mark the severity of pain perceived at rest, during active use, and at night on a 10 cm long horizontal line with the words "0 (no pain)" at the beginning and "10 (most intense pain)" at the end. The individual's pain severity will be recorded by measuring the distance marked on the line in millimeters.
Pressure pain threshold | From baseline to the end of treatment at 10 days
  Pressure pain threshold measurement will be used for digital algometer (Lafayette Manual Muscle Test System ™, Model 01163, Lafayette Instrument Company, Lafayette, In, USA). Before the measurement, all individuals will be informed about the test. During the measurement, individuals will be asked to sit in a comfortable and neutral position in a comfortable and neutral position to come into contact with the soles of the foot. Masseter and temporalis anterior's most swollen, upper trapeze is painful nervous point. The pressure will be applied with a disk head of 1 cm² and the power unit will be set to kg/cm². Values will be recorded by telling the patient to give a "stop" command as soon as he first feels the pain. The averages will be taken twice from the same point.

SECONDARY OUTCOMES:
Range of motion | From baseline to the end of treatment at 10 days
  Cervical flexion, extension, lateral flexion and rotation degrees will be evaluated with universal gonyometer before and after treatment. The ruler will be used to evaluate the maximum oral opening, right left lateral shifts.
The Depression-Anxiety-Stress Scale (DAS) | From baseline to the end of treatment at 10 days
  The Depression-Anxiety-Stress Scale (DAS), developed by Lovibond, was converted into a 21-item short form by Henry and Crawford and adapted to Turkish by Sarıçam (Henry & Crawford, 2005; Lovibond & Lovibond, 1995; Sariçam, 2018). Cronbach's alpha internal consistency reliability coefficient was found to be α=0.87 for the depression subscale, α=0.85 for the anxiety subscale, and α=0.81 for the stress subscale. The 4-point Likert-type scale includes 7 questions to measure depression, stress, and anxiety dimensions, and each section is evaluated within itself. According to the total scores obtained, classification is made as normal, mild, moderate, severe, and very severe.
Insomnia Severity Index (ISI) | From baseline to the end of treatment at 10 days
  It was published by Morin in 1993, and the first psychometric evaluations were published in 2001. The scale, whose Turkish reliability and validity were made by Boysan et al., consists of 7 questions and each item is scored between 0-4. In addition to being a self-reporting tool, the scale is also a tool that can be used by a clinician or another person (e.g. spouse) in evaluation.
Bruxism | From baseline to the end of treatment at 10 days
  It was examined with Bruxism Questionnaire. According to the survey questions prepared by referencing the studies of Pintado et al and Shetty et al, it was stated that individuals who answered "Yes" to at least two of the questions specified in the survey can be called bruxists. The total score range varies between 0-6.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Health Services Vocational School, Bartın, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We can share the questionnaires and indexes used in the study
Supporting Information: Study Protocol